CLINICAL TRIAL: NCT04555538
Title: Atrial Cardiac Magnetic Resonance Imaging in Patients With Embolic Stroke of Unknown Source Without Documented Atrial Fibrillation
Brief Title: Atrial CMR in Patients With CVA of Unknown Source and no Known AF
Acronym: CARM-AF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College Hospital NHS Trust (Other); King's College London (Other); British Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 269654
Record Dates: First submitted 2020-09-14; First posted 2020-09-18 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2020-10

CONDITIONS: Stroke, Ischemic; Atrial Fibrillation
MeSH Terms: conditions — Ischemic Stroke; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Atrial Fibrillation Group
  Interventions: Diagnostic Test: Cardiac MRI
- Non-Atrial Fibrillation Group
  Interventions: Diagnostic Test: Cardiac MRI

INTERVENTIONS:
Diagnostic Test: Cardiac MRI — These are routinely performed for many cardiac conditions, including atrial arrhythmias. The adverse effects are small but include claustrophobia and metallic objects. Therefore all patients will be counselled prior to the scans by an experienced MRI practitioner and standard measures will be taken to avoid distress during the scan. Furthermore, patients will be screened using routine clinical protocols in order to avoid any harm due to interaction of the MRI scanner with metallic objects.

SUMMARY:
This research study will investigate a new method for identifying which patients should be offered blood thinners or therapies to reverse the underlying causes after stroke.

Atrial fibrillation(AF) is the primary risk factor for ischaemic stroke, increasing the risk by up to 5-fold. In AF, the upper heart chambers don't pump blood effectively into the lower chambers. When this happens, a blood clot can form, dislodge and leave the heart blocking an artery in the brain and cause a stroke. However, AF is often an intermittent condition and therefore difficult to diagnose. As such, there are a group of patients in whom no cause of their stroke can be identified.

In this study, we will recruit 92 patients from Guy's and St Thomas' Hospital, Princess Royal University Hospital and King's College London.

As part of routine clinical care, patients undergo insertion of an Implantable Loop Recorder (CE Marked device), a minimally invasive procedure that allows accurate beat-to-beat monitoring to identify patients who develop intermittent AF post-stroke. We will request access to the data collected from this device and perform atrial MRI imaging in these patients to compare the findings between patients that do and do not have AF. If we show that atrial MRI scans are significantly different between patients with and without AF, we will use this information to support a trial of starting appropriate therapies (e.g. blood thinners) in these patients on the basis of MRI findings. This approach would have the advantage of enabling therapies to be offered to the right patients earlier and prevent repeat, potentially disabling stroke.

ELIGIBILITY:
Inclusion Criteria:

Patients will be recruited within 3 months of an acute ischaemic stroke. It must also be feasible to perform a cardiac MRI on all patients enrolled within 3 months of the acute ischaemic stroke.

Inclusion criteria includes patients with:

* Patient consent or advice given by consultee can be obtained
* Confirmed acute ischaemic stroke with evidence on brain CT and/or MRI within 3 months of study enrolment • Ischaemic stroke of unknown source Expected survival >12 months.
* At least one additional stroke risk factor (i.e. CHA2DS2VASc>=3)
* Sinus rhythm on 12 lead ECG, telemetry and a regular pulse on clinical examination
* Above 18 years of age

Exclusion Criteria:

* Unable to obtain patient consent or advice by consultee
* History of atrial fibrillation
* Atrial fibrillation detected on ECG and/or telemetry (AF duration of at least 30 seconds required for diagnosis)
* eGFR <30ml/min
* Indication for pacemaker/implantable cardioverter-defibrillator
* Contra-indication to undergo cardiac MRI (e.g. severe claustrophobia, unable to lie flat for prolonged period, contrast allergy)
* Carotid stenosis >50% on Duplex ultrasound associated with anterior circulation infarction
* Vertebrobasilar stenosis >50% on CT/MR angiography associated with posterior circulation infarction
* Single, isolated lacunar stroke with a corresponding lacunar infarct on brain CT/MRI
* Specific aetiology for cause of stroke (e.g. arteritis, dissection, drug abuse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited during outpatient clinics and inpatient stays
Sampling Method: Non-Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
AF Predictors | 1 year
  Determine if atrial CMR imaging can predict the occurrence of atrial fibrillation in advance of the clinical arrhythmia in patients with confirmed ischaemic stroke

CONTACTS AND LOCATIONS:
Overall Officials: Steven Williams, MBChB PhD, Principal Investigator — King's College London
Locations (3):
- United Kingdom (3):
  - Guy's and St Thomas' Hospital, London
  - King's College Hospital, London
  - Princess Royal University Hospital, Orpington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kotadia ID, O'Dowling R, Aboagye A, Crawley RJ, Bodagh N, Gharaviri A, O'Hare D, Solis-Lemus JA, Roney CH, Sim I, Ramsey D, Newby D, Chiribiri A, Plein S, Sztriha L, Scott P, Masci PG, Harrison J, Williams MC, Birns J, Somerville P, Bhalla A, Niederer S, O'Neill M, Williams SE. High Prevalence of New Clinically Significant Findings in Patients With Embolic Stroke of Unknown Source Evaluated by Cardiac Magnetic Resonance Imaging. J Am Heart Assoc. 2024 Feb 6;13(3):e031489. doi: 10.1161/JAHA.123.031489. Epub 2024 Jan 19. PMID 38240222